CLINICAL TRIAL: NCT02465112
Title: A Randomized Phase III of Adjuvant Targeted Radionuclide Therapy With In111-Pentetreotide in Patients With Digestive Neuroendocrine Tumors After Complete Surgical Resection of Liver Metastases.
Brief Title: Metabolic Radiotherapy After Complete Resection of Liver Metastases in Patient With Digestive Neuroendocrine Tumor
Acronym: TERAVECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Although the relevance of this study remains, the recruitment was too slow (4 patients in 2 years).
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERAVECT D13-2
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Digestive Neuroendocrine Tumors; Metabolic Radiotherapy; Resection; Liver Metastases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metabolic radiotherapy (Experimental): In111-Pentetréotide at 12, 18 and 24 weeks after surgery,
  Interventions: Drug: In111-Pentetréotide
- No metabolic radiotherapy - simple monitoring (Active Comparator): No metabolic radiotherapy - simple monitoring without theraoy
  Interventions: Other: simple monitoring without active therapy

INTERVENTIONS:
Drug: In111-Pentetréotide
  Arms: metabolic radiotherapy
Other: simple monitoring without active therapy
  Arms: No metabolic radiotherapy - simple monitoring

SUMMARY:
TERAVECT is a phase III randomized study of patients with digestive neuroendocrine tumors after complete surgical resection of liver metastases treated with In111-Pentetreotide-based adjuvant radiotherapy.

In this study, targeted radionuclide therapy is used at an earlier stage of the disease.The objective is to target residual tumor cells and/or micrometastases which escaped surgical resection. Given the poor prognosis associated with recurrence, this treatment should prevent relapse.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent,
* Age ≥ 18 years,
* Patients with well differenciated digestive neuroendocrine tumors and liver metastases, for whom a complete surgical resection of liver metastases and of the primary tumor was performed, in 1 or 2 times,
* Immunohistochemical confirmation of neuroendocrine tumors with WHO 2010 grading specification and Ki67 determined of the surgical specimen,
* ECOG Performance Status (PS) 0-1,
* Adequate hematological status: Platelets >100000/mm3, Hemoglobin >10g/dL,
* Adequate Clearance Creatinine >60 mL/min,
* Adequate liver function: Total Serum Bilirubin <1.5x upper limit of normal (ULN), transaminases <3 x ULN,
* Grade of In111-Pentetreotide uptake ≥ 2 (scored according to the Krenning et al scale.: more intense than physiological liver uptake),
* Treatment started within 14 weeks after surgical resection,
* Men and women are required to use adequate birth control measures during the course of the study and for a period of 12 months after the last administration of study drug. Female patients with childbearing potential must have a negative serum pregnant test (β-HCG) within 7 days before starting study treatment,
* Life expectancy >6 months
* Registration with the National Health Care System (CMU included for France)

Exclusion Criteria:

* History of previous or second cancer or progressive cancer occurring within 5 years prior to inclusion, except for basal cell or squamous cell carcinoma,
* Patients with known sensibility or hypersensibility to In111- Pentetreotide or any component of the treatment drug,
* Pregnant or breast-feeding women without adequate birth control measures,
* Patient with known medical history of psychological or psychiatric disorders that may affect patient participation in study due to lack of cooperation or loss of autonomy preventing hospitalization and initiation of study treatment (in good radiation protection conditions),
* Treatment with any investigational drug within 28 days prior to study entry,
* Patient protected by law (tutelage or guardianship).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-09; Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
relapse-free survival (RFS) | up to 3-year

SECONDARY OUTCOMES:
Quality of life (EORTC QLQ-C30) | up to 5-year
  At Baseline, 12, 18 et 24 weeks during therapy, then every 6 months during follow up
Tolerability | up to 5-year after surgery
  Hematological and renal tolerability
Overall survival (1) | up to 3-year
Overall survival (2) | up to 5-year
Identify predictive factors of RFS | Up to 3-year
  Predictive factor : primary tumor location, proliferation index, bilobar or unilobar invasion, number of resected tumors and intratumoral SST2 density immunohistochemical detection.
Impact of the therapy on 1-year RFS in treatment and control group | Up to 1-year
Impact of the therapy on 5-year RFS in treatment and control group | Up to 5-year

CONTACTS AND LOCATIONS:
Overall Officials: Rachida LEBTAHI, MD, Study Director — Hôpital Beaujon
Locations (5):
- France (5):
  - Hôpital Haut Lévêque - CHU Bordeaux, Bordeaux
  - Hôpital Beaujon, Clichy
  - Hôpital R. Salengro, Lille
  - Hôpital Hôtel Dieu, Nantes
  - Hôptal Cochin, Paris